CLINICAL TRIAL: NCT01595243
Title: Effects of Telephone Follow- up Consultations on Discharged Liver Cancer Following Non-surgical Treatment
Brief Title: Effects of Telephone Consultations on Discharged Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 200908011R
Record Dates: First submitted 2012-04-04; First posted 2012-05-10 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Needs; Telephone consultation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): patient with liver cancer in non-surgical treatment after discharge receive usual care
- patient in experiment (Experimental): patient in the experimental group will receive seven instances of telephone follow-up or face to face education
  Interventions: Behavioral: telephone consultations about psychoeducation program

INTERVENTIONS:
Behavioral: telephone consultations about psychoeducation program — experimental group will receive seven instances of telephone follow-up or face-to-face education (the day before discharge and during the first, second, third, fourth, sixth, and eighth weeks after discharge).
  Arms: patient in experiment

SUMMARY:
The aims of this three-year study are to:

1. From patients and family perspective to explore the needs for home care after receiving TACE, PEI, and RFA
2. Develop a telephone follow-up and consultation program and examine its effect on self-efficacy, anxiety, depression and quality of life in liver cancer patients receiving non-surgical treatment.

DETAILED DESCRIPTION:
In the first year, a longitudinal mixed method with quantitative and qualitative method will be used. The Distress Management Tool, the Hospital Anxiety and Depression Scale, and the Short Form-12 quality of life will be used to assess patients' care needs, anxiety, depression, and quality of life in the quantitative method. Data will be analyzed by descriptive, Pearson's Correlation, and Stepwise Regression for each time point. Tape-recorded and in-depth interviews with semi-structured interview guidelines will be used in qualitative method to interview the cancer patients who are scheduled to be discharged after treatment. Content analysis will be used to analyze the interview content.

In the second and third year, randomized control trial will be used to recruit eligible subjects from inpatients in oncology wards in one medical center in Taipei. The eligible subjects will be randomized into a control or experimental group. The patients in the control group will receive usual care and those in the experimental group will receive seven instances of telephone follow-up or face-to-face education (the day before discharge and during the first, second, third, fourth, sixth, and eighth weeks after discharge).Data will be analyzed by independent t-test, one-way analysis of variance, and generalized estimating equations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cancer in non-surgical treatment
* Aged above 18
* Those who are wiling to participate in the research

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
12-Item Short Form Survey | 3 months after discharge
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-ching shun, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan